CLINICAL TRIAL: NCT05269420
Title: Single Anastomosis Sleeve Jejunal Bypass as a Revisional Operation After Restrictive Bariatric Proceures
Brief Title: Single Anastomosis Sleeve Jejunal Bypass as a Revisional Bariatric Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Alaa Mstafa Hassan Sewefy, Assistant professor & consultant of general surgery, Department of Surgery, Minia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ac.med.21.23
Record Dates: First submitted 2022-02-25; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SAS-J (Experimental): single anastomosis sleeve Jejunal Bypass as a revisional bariatric procedure after restrictive bariatric procedures
  Interventions: Procedure: SAS-J

INTERVENTIONS:
Procedure: SAS-J — Single Anastomosis Sleeve Jejunal Bypass

SUMMARY:
single anastomosis sleeve jejunal bypass as a revisional procedure after weight regain or failure after laparoscopic sleeve gastrectomy, gastric plications or laparoscopic adjustable gastric band

DETAILED DESCRIPTION:
in this study the investigators aim to test the efficacy of single anastomosis sleeve jejunal bypass as a revisional procedure after weight regain or failure after laparoscopic sleeve gastrectomy, gastric plications or laparoscopic adjustable gastric band

ELIGIBILITY:
Inclusion Criteria:

obese patients with BMI more than 40 with or without co-morbidity or more than 35 with co-morbidity

* patients fit for laparoscopic surgery
* give approval to share in the study
* previous restrictive bariatric procedure

Exclusion Criteria:

* patients unfit for surgery
* patients aged less than 18 and older than 60
* patient with previous upper abdominal surgery either for obesity or other diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2021-01-04 (Actual)

PRIMARY OUTCOMES:
weight loss | 12 months
  percentage of excess weight loss in kilogram

SECONDARY OUTCOMES:
the rate of improved co morbidity | 12 months
  the effect of the operation on co morbidity like diabetes and hypertension
  the effect of the operation on co morbidity like diabetes and hypertension the effect of single anastomosis sleeve jejunal bypass of comorbidities
the incidence of nutritional deficiency | 12-24 months
  the incidence of nutritional deficiency like anemia, hypocalcamia, hypoproteinemia.
  the incidence of nutritional deficiency like ca, iron, vitaminD and protein malnutrition
the incidence of early operative complications the incidence of early operative complications the incidence of early operative complications the incidence of complications | 12-24 months
  early operative complications like leak, bleeding
  complications like leak, bleeding, dumping,

CONTACTS AND LOCATIONS:
Locations (1):
- Minia university hospital, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided